CLINICAL TRIAL: NCT02023255
Title: A Double-Blind, Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-39393406 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-39393406 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015760; 39393406EDI1002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-39393406; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — JNJ-39393406

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A: Cohort 1 (Experimental): 8 participants will be included in this cohort. 6 participants will receive a single dose of 50 mg JNJ-39393406 and 2 participants will receive placebo for 7 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part A: Cohort 2 (Experimental): 8 participants will be included in this cohort. 6 participants will receive a single dose of 150 mg JNJ-39393406 and 2 participants will receive placebo for 7 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part A: Cohort 3 (Experimental): 8 participants will be included in this cohort. 6 participants will receive a single dose of 450 mg JNJ-39393406 and 2 participants will receive placebo for 7 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part A: Cohort 4 (Experimental): 8 participants will be included in this cohort. 6 participants will receive a single dose of 1,350 mg JNJ-39393406 and 2 participants will receive placebo for 7 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part A: Cohort 5 (Experimental): 8 participants will be included in this cohort. 6 participants will receive a single dose of 2,700 mg JNJ-39393406 and 2 participants will receive placebo for 7 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part B: Cohort A (Experimental): 16 participants will be included in this cohort. 12 participants will receive a single dose of JNJ-39393406 selected based on the pharmacokinetic (PK) data from Part A of the study and 4 participants will receive placebo for 13 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part B: Cohort B (Experimental): 16 participants will be included in this cohort. 12 participants will receive a single dose of JNJ-39393406 selected based on the PK data from Part A of the study and 4 participants will receive placebo for 13 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo
- Part B: Cohort C (Experimental): 16 participants will be included in this cohort. 12 participants will receive a single dose of JNJ-39393406 selected based on the PK data from Part A of the study and 4 participants will receive placebo for 13 consecutive days.
  Interventions: Drug: JNJ-39393406; Other: Placebo

INTERVENTIONS:
Drug: JNJ-39393406 — In Part A of the study, participants will receive single dose of JNJ-39393406 50 mg, 150 mg, 450 mg, 1,350 mg, and 2,700 mg once daily for 7 consecutive days. In Part B of the study, participants will receive single dose of JNJ-39393406 based on the PK data from Part A of the study once daily for 13 consecutive days.
Other: Placebo — In Part A of the study, participants will receive placebo for 7 consecutive days and in Part B of the study, participants will receive placebo for 13 consecutive days.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple dose administration of JNJ-39393406 in young healthy participants, and subsequently in healthy elderly participants.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (study in which an inactive substance is given to one group of participants, while the study medication is given to another group), randomized (the study medication is assigned by chance), and multiple ascending dose (participants will receive multiple doses of study medication and the dose level is subsequently escalated in further groups) study. This study will consist of screening phase (between 21 and 2 days prior to dose administration), a double-blind treatment phase (Part A - 7 days and Part B - 13 days), and a follow-up phase (within 7 to 14 days after last dose administration). In Part A of the multiple ascending dose study approximately 40 young healthy male participants will be randomly allocated to 5 cohorts (group of individuals with similar characteristics) to receive single daily doses of either JNJ-39393406 or placebo for 7 consecutive days. After each dose level, safety, tolerability, and pharmacokinetic (PK) profile (explores what the body does to a medication) of the dose level will be evaluated and the next dose level will be escalated considering the safety and tolerability data. In Part B of the study approximately 48 elderly healthy male and female participants will be randomly allocated to A, B, and C cohorts to receive single daily doses of either JNJ-39393406 or placebo for 13 consecutive days. Dose levels in Part B will be selected based on the PK data from Part A. In both Part A and Part B of the study the dose levels will be increased only after acceptable safety and tolerability data will be obtained. Safety evaluations will include assessments of adverse events, clinical laboratory tests, 24-hour creatinine clearance, Holter monitoring, telemetry, electrocardiogram, vital signs, physical examination, and neurological examination. The study duration for each participant will be approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing to adhere to the prohibitions and restrictions specified in the protocol
* Part A: Body mass index (BMI) between 18 and 30 kg/m2, inclusive (BMI = weight/height2)
* Part B: Female participants must be postmenopausal (for at least 12 months)
* BMI between 18 and 33 kg/m2, inclusive

Exclusion Criteria:

* Clinically significant abnormal values for clinical chemistry, hematology or urinalysis at screening or admission. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening. Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable
* Clinically significant abnormal 24 hour Holter monitoring at screening in the opinion of the investigator
* Significant history of or current psychiatric or neurological illness
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus antibodies at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to Day 56
Maximum Observed Plasma Concentration (Cmax) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Maximum Observed Plasma Concentration (Cmax) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[t]) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  The Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[t]) is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[t]) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  The Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[t]) is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[infinity]) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  The AUC(infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[infinity]) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  The AUC(infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Terminal Rate Constant (Lambda[z]) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  Lambda(z) is defined as terminal rate-constant which reflect the speed of drug elimination in vivo (within the living), and is estimated by log-linear regression analysis of the terminal phase of the plasma concentration versus time curve for at least 3 points.
Terminal Rate Constant (Lambda[z]) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  Lambda(z) is defined as terminal rate-constant which reflect the speed of drug elimination in vivo (within the living), and is estimated by log-linear regression analysis of the terminal phase of the plasma concentration versus time curve for at least 3 points.
Plasma Decay Half-Life (t1/2) of JNJ-39393406 in Part A of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2 to 6 (predose), Day 8 (24 hours), and Days 9, 10 (48/72 hours)
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Plasma Decay Half-Life (t1/2) of JNJ-39393406 in Part B of the study | Days 1 and 7 (predose, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 hours), Days 2, 3, 4, 5, 6, 8, 9, 10, 11, 13 (predose), Day 12 (predose, 1, 2, 4, 6, 8 hours), Day 14 (24 hours), and Days 15, 16 (48/72 hours)
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Change from baseline in cognition in elderly and young healthy participants in Part A of the study | Baseline to Day 6
  For cognitive testing a computerized test battery will be applied, focusing on memory, executive function and attention.
Change from baseline in cognition in elderly and young healthy participants in Part B of the study | Baseline to Day 13
  For cognitive testing a computerized test battery will be applied, focusing on memory, executive function and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium